CLINICAL TRIAL: NCT06752434
Title: Deep Brain Stimulation of the Posterior Subthalamic Area (PSA) Versus Subthalamic Nucleus (STN) for Dystonic Tremor: a Prospective, Randomized, Double-blinded, Cross-over Trial
Brief Title: PSA Versus STN DBS for DT
Acronym: PSA-STN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Suzhou Sceneray Medical Co. , Ltd (Industry); Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, LI DIANYOU, Doctor, Ruijin Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DTPSASTN
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Dystonic Tremor
Keywords: Dystonic Tremor; deep brain stimulation; posterior subthalamic area; subthalamic nucleus
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSA-STN (Experimental): Participants randomized in this arm will receive bilateral PSA stimulation in the first two months in the randomized phase and then will be crossovered to the bilateral STN stimulation for another two months.
  Interventions: Device: Deep brain stimulation
- STN-PSA (Experimental): Participants randomized in this arm will receive bilateral STN stimulation in the first two months in the randomized phase and then will be crossovered to the bilateral PSA stimulation for another two months.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — active DBS with optimal stimulating parameters

SUMMARY:
The aim of this study is to compare the effectiveness of the deep brain stimulation in the posterior subthalamic area (PSA) versus the subthalamic nucleus (STN) for the treatment of dystonic tremor (DT) in a randomized, double-blinded, cross-over manner.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, crossover trial aiming at comparing the efficacy of PSA and STN DBS in treating dystonic tremor. Enrolled patients will undergo bilateral DBS surgery, targeting both PSA and STN with single trajectory. Three months post-implantation, patients enter a 4-month double-blinded crossover phase with PSA and STN DBS in randomized order. After 7 months post-implantation (at the end of the crossover phase), patients enter an open-label phase during which programming parameters are not restricted until the termination of the study at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dystonic tremor based on the MDS 2018 consensus
* Duration of DT symptoms: ≥3 years of motor symptoms
* If the patient is taking tremor medications, the medications should be stable for 28 days prior to informed consent
* Good compliance and written informed consent

Exclusion Criteria:

* Any intracranial abnormalities that would prevent DBS surgery
* Any significant mental illness that might affect the subject's ability to comply with the study protocol requirements (e.g., bipolar disorder, schizophrenia, mood disorders with psychotic features, Cluster B personality disorders)
* Severe cognitive impairment, MOCA score <24
* Any current substance or alcohol abuse according to DSM-V criteria
* Any history of recurrent or unprovoked epileptic seizures; any prior movement disorder treatment involving intracranial surgery or device implantation; any history of hemorrhagic stroke; any significant medical condition that might interfere with the study procedures or could confound the assessment of study endpoints
* Any terminal illness with a life expectancy of <1 year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Fahn-Tolosa-Marin Clinical Rating Scale for Tremor to 5 months | 5 months
Change from baseline Fahn-Tolosa-Marin Clinical Rating Scale for Tremor to 7 months | 7 months

SECONDARY OUTCOMES:
Change from baseline Burke-Fahn-Marsden Dystonia Rating Scale to 5 months | 5 months
Change from baseline Burke-Fahn-Marsden Dystonia Rating Scale to 7 months | 7 months
Change from baseline Mini-Mental Status Exam to 5 months | 5 months
Change from baseline Mini-Mental Status Exam to 7 months | 7 months
Change from baseline Beck depression inventory to 5 months | 5 months
Change from baseline Beck depression inventory to 7 months | 7 months
Adverse events | up to 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dianyou Li, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China